CLINICAL TRIAL: NCT01050933
Title: Safety and Tolerability of Inhaled Carbon Monoxide in Healthy Volunteers
Brief Title: Safety Study of Inhaling Carbon Monoxide in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: resident left and no one to take over
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Paul Belliveau, Principal Investigator, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POICO-A
Record Dates: First submitted 2010-01-13; First posted 2010-01-18 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Healthy volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carbon Monoxide (Experimental): Healthy volunteers will receive 250 ppm of carbon monoxide by face mask. This dose will be administered for 1 hour with continuous COHb monitoring. At baseline and at each half hour time point, a blood sample will be drawn to be analyzed by the gas chromatograph. After 1 hour, the volunteer will be excused and asked to return in 4 hours and this procedure repeated. At any point, if the COHb level reaches 10%, administration of CO will be terminated.
  Interventions: Drug: 250 ppm carbon monoxide

INTERVENTIONS:
Drug: 250 ppm carbon monoxide — 250 ppm of inhaled carbon monoxide over one hour

SUMMARY:
Post operative ileus (POI), a temporary paralysis of the intestines, is a serious health care problem. It normally occurs in all patients after surgery to the abdomen but in some cases can result in serious complications. The objective of this study is to determine if inhaling very low doses of carbon monoxide (CO) before and after colon surgery will shorten the duration of normal POI and/or prevent the development of POI complications in patients undergoing colon surgery.

This preliminary study will be conducted in ten healthy volunteers to monitor for blood levels and adverse effects that occur at different durations of exposure of inhaled CO to establish a safe dose for patients in the main trial. For the main trial, patients requiring surgery to their colon will be assigned randomly to receive one hour treatments of either CO or oxygen by face mask before and after their operation.

We hypothesize that healthy volunteers will be able to tolerate 1 hour doses of 250 ppm of CO with minimal side effects. It is also anticipated that for each dose of CO administered, the blood levels of CO will remain well under poisonous levels. Finally, we anticipate blood levels of CO will return to baseline level within 24 hours following the last dose of CO.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age > 18 years.
* Women must be using acceptable contraceptives, post-menopausal or surgically sterile.
* No prior smoking history.
* BMI between 16 and 30 inclusive.
* In good health as per medical history, physical exam, vital signs & ECG.

Exclusion Criteria:

* Exposure to carbon monoxide during the 48 hours prior to the study day.
* Occupational exposure to CO.
* Significant disease that may put the volunteer at risk because of participation in the study or may influence the results of the study or the volunteer's ability to participate in the study.
* Baseline blood level of COHb >2%.
* Patients with underlying lung disease such as asthma or COPD.
* Baseline oxygen saturation <92% on room air.
* Planned pregnancy, already pregnant or breastfeeding.
* Participation in another clinical trial within 2 months prior to study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Adverse Event Rate | Before and after carbon monoxide exposure

CONTACTS AND LOCATIONS:
Overall Officials: Paul Belliveau, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada